CLINICAL TRIAL: NCT02737904
Title: The Effect of Cycling Using Active-passive Trainers on Spasticity, Cardiovascular Fitness, Function and Quality of Life in People With Multiple Sclerosis
Brief Title: Effect of Active-Passive Trainer Cycling on Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GN15PY148; PRF-15-BO1 (Other Grant/Funding Number: Chartered Society of Physiotherapy Charitable Trust Award)
Record Dates: First submitted 2016-04-04; First posted 2016-04-14 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Multiple Sclerosis
Keywords: Muscle spasticity
MeSH Terms: conditions — Multiple Sclerosis; Muscle Spasticity | interventions — APT

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Active Comparator): Usual care - conventional, personalised in-patient rehabilitation 4 weeks duration
  Interventions: Other: Usual care
- Intervention group (Experimental): Usual care - conventional, personalised in-patient rehabilitation - plus APT cycling programme 4 weeks duration
  Interventions: Other: APT; Other: Usual care

INTERVENTIONS:
Other: APT — APT for 30 minutes per day on 5 days per week for 4 weeks: 2 minute warm up consisting of passive cycling, where the legs of the participant are moved passively by the APT at 10 revolutions per min (rpm). Next, the participant will cycle for up to 26 minutes, at 60rpm. In this phase, the participant is required to actively cycle and to maintain a symmetrical pattern of movement using the feedback on the display. If the participant is unable to actively cycle at any point during the 26 minute exercise period, or if they have a spasm, the MOTOmed APT will revert to the passive mode. The final phase is a cool down where participants again will have 2 minutes of passive cycling at 10rpm.
  Arms: Intervention group
Other: Usual care — Personalised in-patient rehabilitation programme

SUMMARY:
This randomised controlled trial aims to explore the effectiveness of a four week programme of exercise using lower limb Active Passive trainer (APT) (MOTOmed trainer) in terms of spasticity in people with moderate to severe Multiple Sclerosis.

DETAILED DESCRIPTION:
Exercise is beneficial for people with Multiple Sclerosis (pwMS). However, exercise options for those with moderate to high levels of disability are limited. Cycling, delivered with an Active Passive Trainer (APT) is one exercise option often offered within rehabilitation/exercise settings and many pwMS buy APTs for home use. Anecdotally, pwMS report they feel better and their spasticity reduces after APT cycling, however there is a lack of evidence to support this.

30 pwMS will be recruited from the Physical Disability Rehabilitation Unit at the Queen Elizabeth University Hospital, Glasgow, and randomised to APT + usual care or usual care only. Those in the APT group will receive 30 minutes of APT (2 mins passive warm up, 26 mins active cycling and 2 mins passive cool down), five days per week for 4 weeks. Outcome measures will be cardiovascular fitness measured using the oxygen uptake efficiency slope (OUES), spasticity assessed by Modified Ashworth Scale (MAS) and the Multiple Sclerosis Spasticity Scale (MSSS-88), function assessed by the Functional Independence Measure (FIM) and the Timed 25 foot walk test (T25FW), Quality of Life measured by MSQOL-54. Outcome measures will be assessed in both groups before and after the 4 week intervention period. Symmetry, distance cycled and power will be recorded following each cycling session in the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* have a confirmed diagnosis of progressive MS
* are aged over 18 years
* have an Expanded Disability Status Scale (EDSS) of between 6.5 (requires two walking aids - pair of canes, crutches, etc - to walk about 20m without resting) and 8.5 (essentially restricted to bed much of day); has some effective use of arms (retains some self care functions) and spasticity in their lower limbs (self reported)

Exclusion Criteria:

* cognitive impairment (cannot understand instructions)
* other co-morbidities which would preclude them taking part in exercise
* visual impairment (such that they cannot see the screen on the APT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Effect of spasticity on daily life scored on Multiple Sclerosis Spasticity Scale (MSSS-88) | Change from Baseline at 4 weeks
  Score on Multiple Sclerosis Spasticity Scale (MSSS-88)

SECONDARY OUTCOMES:
Spasticity scored on Modified Ashworth Scale (MAS) | Change from Baseline at 4 weeks
  Score on Modified Ashworth Scale (MAS)
Cardiovascular fitness calculated using Oxygen Uptake Efficiency Slope (OUES) | Change from Baseline at 4 weeks
  Calculated Oxygen Uptake Efficiency Slope (OUES)
Function - FIM | Change from Baseline at 4 weeks
  Score on Functional Independence Measure (FIM)
Function - T25FW | Change from Baseline at 4 weeks
  Timed 25-foot walk test (T25FW)
Quality of Life (MSQOL)-54 scale | Change from Baseline at 4 weeks
  Score on Multiple Sclerosis Quality of Life (MSQOL)-54 scale
APT cycling performance - symmetry | Change from Baseline at 4 weeks
  Proportion of time when effort of right versus left leg is evenly distributed ie 50%/50%
APT cycling performance - distance | Change from Baseline at 4 weeks
  Distance cycled
APT cycling performance - power | Change from Baseline at 4 weeks
  Overall power (measured in watts)

CONTACTS AND LOCATIONS:
Overall Officials: Lorna Paul, BSc MPhil PhD, Principal Investigator — University of Glasgow
Locations (1):
- Physical Disability Rehabilitation Unit (PDRU), Queen Elizabeth University Hospital, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No